CLINICAL TRIAL: NCT06169384
Title: Endoscopic Partial Adenoidectomy Versus Total Adenoidectomy Regarding Rate of Recurrence and Relief of Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Mahmoud Mohamed Ragheb, Resident investigator, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Endoscopic adenoidectomy
Record Dates: First submitted 2023-11-28; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Adenoidal Hypertrophy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic total adenoidectomy (Active Comparator)
  Interventions: Device: Endoscopic adenoidectomy
- Endoscopic partial adenoidectomy (Active Comparator)
  Interventions: Device: Endoscopic adenoidectomy

INTERVENTIONS:
Device: Endoscopic adenoidectomy — Subjects will be randomly assigned into two groups (30 patient each group): Group A will undergo endoscopic partial adenoidectomy using the 70◦ rigid endoscope trans-orally and shaver (microdebrider) ,by removing the upper (choanal) part only with leaving the lower part of the adenoid .(2) Group B will undergo total adenoidectomy ,by removing all the adenoid lymphoid tissue .

SUMMARY:
Efficacy of partial adenoidectomy versus total adenoidectomy regarding rate of recurrence and relief of nasal obstruction.

ELIGIBILITY:
Inclusion Criteria:

* .all patients with adenoid hypertrophy causing airway obstruction.

Exclusion Criteria:

* 1. Chlidren known to have cleft palate ,submucous cleft palate or other medical problems causing velopharyngeal insufficiency.
* 2 . Systemic medical problems interfering with surgery.
* 3 . Refusal of parents to participate.
* 4. Craniofacial abnormalities.
* 5. Down syndrome.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of partial adenoidectomy versus total adenoidectomy regarding rate of recurrence and relief of nasal obstruction. | 1 to 2 years .
  1. Relief of nasal obstruction while preserving the function of velopharyngeal valve and assessment of the recurrence rate.
Incidence of recurrence using fibro-optic evaluation | 1 to 2 years .
  Relief of nasal obstruction of posterior nasal chona using fibro-optic evaluation and assessment of recurrence rate using also questionnaires sheets to all parents.

CONTACTS AND LOCATIONS:
Locations (1):
- AssiutU, Asyut, Egypt

REFERENCES:
- [Background] 1. Jervis-Bardy, J.; Department of Otolaryngology, Arkansas Children's Hospital, cLittle Rock, AR, United States. Journal of Craniofacial SurgeryVolume 30, Issue 5, Pages E454 - E4602019.
- [Background] 1. Kummer AW, Lee L. Evaluation and treatment of resonance disorders. Language, Speech, and Hearing Services in Schools, 27:271-281
- [Background] Saunders NC, Hartley BE, Sell D, Sommerlad B. Velopharyngeal insufficiency following adenoidectomy. Clin Otolaryngol Allied Sci. 2004 Dec;29(6):686-8. doi: 10.1111/j.1365-2273.2004.00870.x. PMID 15533160